CLINICAL TRIAL: NCT04617275
Title: A 12-WEEK, PHASE 2A, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, PARALLEL GROUP STUDY TO ASSESS THE SAFETY, TOLERABILITY, AND PHARMACODYNAMICS OF PF-06882961 TITRATION IN ADULTS WITH TYPE 2 DIABETES MELLITUS TREATED WITH METFORMIN AND IN NON-DIABETIC ADULTS WITH OBESITY
Brief Title: A 12-WEEK TITRATE STUDY TO EVALUATE SAFETY, TOLERABILITY AND PHARMACODYNAMICS OF PF-06882961 IN ADULTS WITH TYPE 2 DIABETES MELLITUS AND IN NON-DIABETIC ADULTS WITH OBESITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C3421008; GLP-1Ra Ph 2 Titration Study (Other: Alias Study Number)
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Results first posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — danuglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm 1-PF-06882961 starting dose of 5 milligram (mg) BID titrated to 120 mg in participants with T2DM (Experimental): The dose will be titrated over 12 weeks, starting with a dose of 5 mg BID to reach the target dose of 120 mg BID. Titration steps include: 5 mg BID, 10 mg BID, 20 mg BID, 40 mg BID, 60 mg BID, 80 mg BID, 100 mg BID and 120 mg BID
  Interventions: Drug: PF-06882961
- Arm 2-PF-06882961 starting dose of 10 mg BID titrated to 100 mg in participants with T2DM (Experimental): The dose will be titrated over 12 weeks, starting with a dose of 10 mg BID to reach the target dose of 120 mg BID. Titration steps include: 10 mg BID, 20 mg BID, 40 mg BID, 60 mg BID, 80 mg BID, 100 mg BID and 120 mg BID
  Interventions: Drug: PF-06882961
- Arm 3-PF-06882961 starting dose of 5 mg BID titrated to 80 mg in participants with T2DM (Experimental): The dose will be titrated over 12 weeks, starting with a dose of 5 mg BID to reach the target dose of 80 mg BID. Titration steps include: 5 mg BID, 10 mg BID, 20 mg BID, 40 mg BID, 60 mg BID and 80 mg BID
  Interventions: Drug: PF-06882961
- Arm 4-PF-06882961 starting dose of 10 mg BID titrated to 80 mg in participants with T2DM (Experimental): The dose will be titrated over 12 weeks, starting with a dose of 10 mg BID to reach the target dose of 80 mg BID. Titration steps include: 10 mg BID, 20 mg BID, 40 mg BID, 60 mg BID and 80 mg BID
  Interventions: Drug: PF-06882961
- Arm 5 - Placebo in subjects with T2DM and Obesity (Placebo Comparator): Matching Placebo tablets taken twice a day (BID)
  Interventions: Other: Placebo
- Arm 6-PF-06882961 starting dose of 10 mg BID titrated to 200 mg in participants with T2DM (Experimental): The dose will be titrated over 12 weeks, starting with a dose of 10 mg BID to reach the target dose of 200 mg BID. Titration steps include: 10 mg BID, 20 mg BID, 40 mg BID, 60 mg BID, 80 mg BID, 100 mg BID and 120 mg BID,140 mg BID, 160 mg BID, 180 MG BID, 200 mg BID
  Interventions: Drug: PF-06882961
- Arm 7-PF-06882961 starting dose of 10 mg BID titrated to 200 mg in participants with Obesity (Experimental): The dose will be titrated over 12 weeks, starting with a dose of 10 mg BID to reach the target dose of 200 mg BID. Titration steps include: 10 mg BID, 20 mg BID, 40 mg BID, 60 mg BID, 80 mg BID, 100 mg BID and 120 mg BID,140 mg BID, 160 mg BID, 180 MG BID, 200 mg BID
  Interventions: Drug: PF-06882961

INTERVENTIONS:
Drug: PF-06882961 — PF-68882961 will be provided as tablets twice a day (BID)
  Arms: Arm 1-PF-06882961 starting dose of 5 milligram (mg) BID titrated to 120 mg in participants with T2DM; Arm 2-PF-06882961 starting dose of 10 mg BID titrated to 100 mg in participants with T2DM; Arm 3-PF-06882961 starting dose of 5 mg BID titrated to 80 mg in participants with T2DM; Arm 4-PF-06882961 starting dose of 10 mg BID titrated to 80 mg in participants with T2DM; Arm 6-PF-06882961 starting dose of 10 mg BID titrated to 200 mg in participants with T2DM; Arm 7-PF-06882961 starting dose of 10 mg BID titrated to 200 mg in participants with Obesity
Other: Placebo — Placebo comparator will be provided as tablets twice daily for 12 weeks
  Arms: Arm 5 - Placebo in subjects with T2DM and Obesity

SUMMARY:
This study will assess tolerability, safety, and pharmacodynamics (PD) of twice daily (BID) administration of PF- 06882961 in adult participants with Type 2 Diabetes Mellitus (T2DM) who are treated with metformin and in non-diabetic adults with obesity

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between the ages of 18 and 75 years, inclusive, at Visit 1 (screening).

Exclusion Criteria:

* Diagnosis of type 1 diabetes mellitus or secondary forms of diabetes.
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, New York Heart Association Functional Class II IV heart failure, or transient ischemic attack within 6 months of screening (Visit 1).
* Participants with a known medical history of active liver disease (other than non alcoholic hepatic steatosis), including chronic active hepatitis B or C, or primary biliary cirrhosis.
* History of major depressive disorder or history of other severe psychiatric disorders (eg, schizophrenia or bipolar disorder) within the last 2 years.
* Any lifetime history of a suicide attempt.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (38):
  - Arizona Research Center, Phoenix, Arizona
  - Unity Health - Searcy Medical Center, Searcy, Arkansas
  - Catalina Research Institute, LLC, Montclair, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - California Research Foundation, San Diego, California
  - University Clinical Investigators, Inc., Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Pines Care Research Center, LLC, Pembroke Pines, Florida
  - Solaris Clinical Research, Meridian, Idaho
  - Meridian Clinical Research, LLC, Sioux City, Iowa
  - Research Integrity, LLC, Owensboro, Kentucky
  - Nola Care LLC, Metairie, Louisiana
  - Clinical Research Professionals, Chesterfield, Missouri
  - Meridian Clinical Research, LLC DBA Regional Clinical Research, Endwell, New York
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - PMG Research of Rocky Mount, LLC - Investigational Product and Mail delivery, Rocky Mount, North Carolina
  - PMG Research of Rocky Mount, LLC - Patient Visits, Rocky Mount, North Carolina
  - Carolina Research Center, Inc., Shelby, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Palmetto Clinical Research, Summerville, South Carolina
  - Palmetto Primary Care Physicians (physicals only), Summerville, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Dallas Diabetes Research Center, Dallas, Texas
  - Juno Research, LLC, Houston, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Bountiful Internal Medicine, Bountiful, Utah
  - Progressive Clinical Research, Bountiful, Utah
  - Wade Family Medicine, Bountiful, Utah
  - Manassas Clinical Research Center, Manassas, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Saxena AR, Frias JP, Gorman DN, Lopez RN, Andrawis N, Tsamandouras N, Birnbaum MJ. Tolerability, safety and pharmacodynamics of oral, small-molecule glucagon-like peptide-1 receptor agonist danuglipron for type 2 diabetes: A 12-week, randomized, placebo-controlled, Phase 2 study comparing different dose-escalation schemes. Diabetes Obes Metab. 2023 Oct;25(10):2805-2814. doi: 10.1111/dom.15168. Epub 2023 Jun 13. PMID 37311722
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 06 January 2021 to 17 November 2021 in the United States.
Pre-assignment Details: A total of 370 participants were screened for eligibility, of which 151 participants (123 in the type 2 diabetes mellitus [T2DM] arms and 28 in the non-diabetic obesity arms) were randomized to receive the danuglipron or placebo in one of the 8 treatment arms.
Groups:
- Placebo (T2DM): Participants with T2DM received matching placebo tablets orally twice daily (BID) with food.
- PF-06882961 80 mg BID Low, Slow (T2DM): Participants with T2DM received PF-06882961 tablets orally BID with food. The dose were titrated from 5 mg to 80 mg over 12 weeks in following steps: 5 mg BID, 10 mg BID, 20 mg BID, 40 mg BID, 60 mg BID and 80 mg BID.
- PF-06882961 80 mg BID High, Slow (T2DM): Participants with T2DM received PF-06882961 tablets orally BID with food. The dose were titrated from 10 mg to 80 mg over 12 weeks in following steps: 10 mg BID, 20 mg BID, 40 mg BID, 60 mg BID and 80 mg BID.
- PF-06882961 120 mg BID Low, Fast (T2DM): Participants with T2DM received PF-06882961 tablets orally BID with food. The dose were titrated from 5 mg to 120 mg over 12 weeks in following steps: 5 mg BID, 10 mg BID, 20 mg BID, 40 mg BID, 60 mg BID, 80 mg BID, 100 mg BID and 120 mg BID.
- PF-06882961 120 mg BID High, Fast (T2DM): Participants with T2DM received PF-06882961 tablets orally BID with food. The dose were titrated from 10 mg to 120 mg over 12 weeks in following steps: 10 mg BID, 20 mg BID, 40 mg BID, 60 mg BID, 80 mg BID, 100 mg BID and 120 mg BID.
- PF-06882961 200 mg BID (T2DM): Participants with T2DM received PF-06882961 tablets orally BID with food. The dose were titrated from 10 mg to 200 mg over 12 weeks in following steps: 10 mg BID, 20 mg BID, 40 mg BID, 60 mg BID, 80 mg BID, 100 mg BID and 120 mg BID,140 mg BID, 160 mg BID, 180 mg BID, 200 mg BID.
- Placebo (Non-diabetic Obesity): Participants with non-diabetic obesity received matching placebo tablets orally BID with food.
- PF-06882961 200 mg BID (Non-diabetic Obesity): Participants with non-diabetic obesity received PF-06882961 tablets orally BID with food. The dose were titrated from 10 mg to 200 mg over 12 weeks in following steps: 10 mg BID, 20 mg BID, 40 mg BID, 60 mg BID, 80 mg BID, 100 mg BID and 120 mg BID,140 mg BID, 160 mg BID, 180 mg BID, 200 mg BID.
Period: Treatment Period
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM) | Placebo (Non-diabetic Obesity) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Started | 16 | 20 | 22 | 22 | 22 | 21 | 6 | 22
Completed | 13 | 13 | 16 | 13 | 13 | 10 | 5 | 6
Not Completed | 3 | 7 | 6 | 9 | 9 | 11 | 1 | 16
Not completed — Adverse Event | 1 | 6 | 4 | 6 | 7 | 8 | 0 | 12
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 2
Not completed — No longer meets eligibility criteria | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 2 | 2 | 0 | 1 | 2
Period: Follow-up Period
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM) | Placebo (Non-diabetic Obesity) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Started | 16 | 20 | 22 | 22 | 22 | 21 | 6 | 22
Completed | 13 | 17 | 18 | 16 | 16 | 14 | 5 | 14
Not Completed | 3 | 3 | 4 | 6 | 6 | 7 | 1 | 8
Not completed — Adverse Event | 1 | 1 | 2 | 3 | 4 | 3 | 0 | 3
Not completed — Lost to Follow-up | 0 | 1 | 2 | 0 | 0 | 4 | 0 | 3
Not completed — No longer meets eligibility criteria | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 2 | 2 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: A total of 151 participants were assigned to the treatment and treated with danuglipron or placebo.
Groups:
- PF-06882961 80 mg BID Low, Slow (T2DM): Participants with T2DM received PF-06882961 tablets orally BID with food. The dose were titrated from 5 mg to 80 mg over 12 weeks.
- PF-06882961 80 mg BID High, Slow (T2DM): Participants with T2DM received PF-06882961 tablets orally BID with food. The dose were titrated from 10 mg to 80 mg over 12 weeks.
- PF-06882961 120 mg BID Low, Fast (T2DM): Participants with T2DM received PF-06882961 tablets orally BID with food. The dose were titrated from 5 mg to 120 mg over 12 weeks.
- PF-06882961 120 mg BID High, Fast (T2DM): Participants with T2DM received PF-06882961 tablets orally BID with food. The dose were titrated from 10 mg to 120 mg over 12 weeks.
- PF-06882961 200 mg BID (T2DM): Participants with T2DM received PF-06882961 tablets orally BID with food. The dose were titrated from 10 mg to 200 mg over 12 weeks.
- PF-06882961 200 mg BID (Non-diabetic Obesity): Participants with non-diabetic obesity received PF-06882961 tablets orally BID with food. The dose were titrated from 10 mg to 200 mg over 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo (T2DM) | Placebo (Non-diabetic Obesity) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM) | PF-06882961 200 mg BID (Non-diabetic Obesity) | Total
Number analyzed (Participants) | 16 | 6 | 20 | 22 | 22 | 22 | 21 | 22 | 151
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean (SD) | 53.9 (9.10) | 49.5 (5.79) | 59.5 (9.55) | 60.9 (8.69) | 58.3 (7.11) | 57.2 (11.8) | 59 (9.31) | 48.5 (13.12) | 56.5 (10.55)
Age, Continuous [Median (Full Range); unit: Years] | 53.0 [39 to 69] | 49.0 [42 to 59] | 60.5 [34 to 72] | 61.5 [46 to 74] | 58.5 [41 to 71] | 60.0 [32 to 75] | 59.0 [44 to 75] | 52.0 [21 to 69] | 58.0 [21 to 75]
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-44 | 2 | 1 | 1 | 0 | 1 | 3 | 1 | 7 | 16
  45-64 | 12 | 5 | 12 | 13 | 18 | 12 | 14 | 13 | 99
  >=65 | 2 | 0 | 7 | 9 | 3 | 7 | 6 | 2 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 10 | 10 | 10 | 10 | 10 | 16 | 78
  Male | 8 | 2 | 10 | 12 | 12 | 12 | 11 | 6 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 6 | 17 | 19 | 19 | 17 | 17 | 18 | 125
  Black or African American | 4 | 0 | 3 | 2 | 2 | 5 | 3 | 4 | 23
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Not reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 9 | 3 | 12 | 11 | 9 | 11 | 15 | 13 | 83
  Not Hispanic or Latino | 7 | 3 | 8 | 11 | 13 | 11 | 6 | 9 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were events between first dose of study drug and up to follow-up visit that were absent before treatment or that worsened after treatment. AEs presented below were TEAEs. The investigator was required to use clinical judgment to assess the potential relationship between investigational product and each AE, to define an treatment-related AE. Assessments of AE intensity were defined as mild (easily tolerated, causing minimal discomfort and not interfering with daily activities), moderate (causing sufficient discomfort and interferes with normal daily activities) and severe (preventing normal daily activities).
Time Frame: Baseline through follow-up (Day 112)
Population: Safety analysis set included all participants randomly assigned to study treatment and who took at least 1 dose of investigational products (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM) | Placebo (Non-diabetic Obesity) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21 | 6 | 22
Participants
  All Causality - Mild | 5 | 4 | 10 | 9 | 8 | 10 | 1 | 6
  All Causality - Moderate | 3 | 8 | 3 | 5 | 6 | 3 | 3 | 11
  All Causality - Severe | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1
  Treatment Related - Mild | 2 | 4 | 8 | 3 | 7 | 9 | 0 | 5
  Treatment Related - Moderate | 2 | 4 | 2 | 3 | 7 | 3 | 1 | 11
  Treatment Related - Severe | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1

2. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Safety laboratory assessments included clinical chemistry, hematology, urinalysis, and other tests. Abnormality was determined at the investigator's discretion.
Time Frame: Baseline through Visit 10 (Day 91)
Population: Safety analysis set included all participants randomly assigned to study treatment and who took at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM) | Placebo (Non-diabetic Obesity) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Number analyzed (Participants) | 15 | 20 | 21 | 21 | 22 | 19 | 6 | 22
Participants | 12 | 16 | 17 | 20 | 17 | 14 | 4 | 9

3. Secondary Outcome: Number of Participants With Vital Signs Meeting the Pre-defined Categorical Summarization Criteria
Description: Vital signs abnormality criteria: 1) supine systolic blood pressure (SBP) <90 millimeters of mercury (mmHg); 2) supine diastolic blood pressure (DBP) <50 mmHg; 3) supine pulse rate <40 or >120 beats per minute (bpm); 4) change from baseline (increase or decrease) in supine SBP >=30 mmHg; 5) change from baseline (increase or decrease) in supine DBP >=20 mmHg.
Time Frame: Baseline through Visit 10 (Day 91)
Population: Safety analysis set included all participants randomly assigned to study treatment and who took at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM) | Placebo (Non-diabetic Obesity) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21 | 6 | 22
Participants
  Supine SBP <90 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine SBP Increase >=30 mmHg | 0 | 0 | 2 | 0 | 4 | 1 | 0 | 0
  Supine SBP Decrease >=30 mmHg | 0 | 2 | 1 | 3 | 2 | 1 | 1 | 2
  Supine DBP <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine DBP Increase >=20 mmHg | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 0
  Supine DBP Decrease >=20 mmHg | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Supine Pulse Rate <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine Pulse Rate >120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting the Pre-defined Categorical Summarization Criteria
Description: ECG assessments included pulse rate (PR), QT, heart rate, QTcF intervals and QRS complex. ECG abnormalities criteria included: PR interval value >= 300 msec, or baseline (BL) >200 msec and >=25% increase from BL, or BL <=200 msec and >=50% increase from BL; QRS interval value >= 140msec, or >=50% increase from BL; QTcF value >450 and <=480 msec, or >480 and <=500 msec, or >500 msec, or increase from BL>30 and <=60 msec, or >60msec.
Time Frame: Baseline through Visit 10 (Day 91)
Population: Safety analysis set included all participants randomly assigned to study treatment and who took at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM) | Placebo (Non-diabetic Obesity) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21 | 6 | 22
Participants
  PR interval >=300 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  %Change in PR interval >=25/50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS interval >=140 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  %Change in QRS interval >=50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval >450 and <=480 msec | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1
  QTcF interval >480 and <=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  QTcF interval >500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change in QTcF interval >30 and <=60 msec | 2 | 0 | 0 | 1 | 3 | 0 | 0 | 0
  Change in QTcF interval >60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

5. Secondary Outcome: Number of Participants With Categorical Scores on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. Participants who responded "yes" to the questions will be counted. Data relevant to the assessment of suicidality were mapped to the Columbia-Classification Algorithm of Suicide Assessment (C-CASA) codes.
Time Frame: Week 0, 2, 4, 6, 8, 10, 12, 13-14
Population: Safety analysis set included all participants randomly assigned to study treatment and who took at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (T2DM) | Placebo (Non-diabetic Obesity) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Number analyzed (Participants) | 16 | 6 | 20 | 22 | 22 | 22 | 21 | 22
Participants
  Week 0 - <1> Completed Suicide: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - <1> Completed Suicide | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - <2> Suicide Attempt: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - <2> Suicide Attempt | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - <3> Preparatory Acts Towards Imminent Suicidal Behavior: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - <3> Preparatory Acts Towards Imminent Suicidal Behavior | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - <4> Suicidal Ideation: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - <4> Suicidal Ideation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - <7> Self-injurious Behavior, No Suicidal Intent: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - <7> Self-injurious Behavior, No Suicidal Intent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - <1> Completed Suicide: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - <1> Completed Suicide | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - <2> Suicide Attempt: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - <2> Suicide Attempt | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - <3> Preparatory Acts Towards Imminent Suicidal Behavior: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - <3> Preparatory Acts Towards Imminent Suicidal Behavior | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - <4> Suicidal Ideation: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - <4> Suicidal Ideation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - <7> Self-injurious Behavior, No Suicidal Intent: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - <7> Self-injurious Behavior, No Suicidal Intent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - <1> Completed Suicide: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - <1> Completed Suicide | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - <2> Suicide Attempt: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - <2> Suicide Attempt | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - <3> Preparatory Acts Towards Imminent Suicidal Behavior: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - <3> Preparatory Acts Towards Imminent Suicidal Behavior | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - <4> Suicidal Ideation: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - <4> Suicidal Ideation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - <7> Self-injurious Behavior, No Suicidal Intent: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - <7> Self-injurious Behavior, No Suicidal Intent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 - <1> Completed Suicide: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 - <1> Completed Suicide | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 - <2> Suicide Attempt: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 - <2> Suicide Attempt | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 - <3> Preparatory Acts Towards Imminent Suicidal Behavior: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 - <3> Preparatory Acts Towards Imminent Suicidal Behavior | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 - <4> Suicidal Ideation: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 - <4> Suicidal Ideation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 - <7> Self-injurious Behavior, No Suicidal Intent: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 - <7> Self-injurious Behavior, No Suicidal Intent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - <1> Completed Suicide: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - <1> Completed Suicide | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - <2> Suicide Attempt: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - <2> Suicide Attempt | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - <3> Preparatory Acts Towards Imminent Suicidal Behavior: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - <3> Preparatory Acts Towards Imminent Suicidal Behavior | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - <4> Suicidal Ideation: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - <4> Suicidal Ideation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - <7> Self-injurious Behavior, No Suicidal Intent: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - <7> Self-injurious Behavior, No Suicidal Intent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - <1> Completed Suicide: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - <1> Completed Suicide | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - <2> Suicide Attempt: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - <2> Suicide Attempt | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - <3> Preparatory Acts Towards Imminent Suicidal Behavior: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - <3> Preparatory Acts Towards Imminent Suicidal Behavior | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - <4> Suicidal Ideation: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - <4> Suicidal Ideation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - <7> Self-injurious Behavior, No Suicidal Intent: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - <7> Self-injurious Behavior, No Suicidal Intent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - <1> Completed Suicide: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - <1> Completed Suicide | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - <2> Suicide Attempt: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - <2> Suicide Attempt | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - <3> Preparatory Acts Towards Imminent Suicidal Behavior: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - <3> Preparatory Acts Towards Imminent Suicidal Behavior | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - <4> Suicidal Ideation: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - <4> Suicidal Ideation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - <7> Self-injurious Behavior, No Suicidal Intent: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - <7> Self-injurious Behavior, No Suicidal Intent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - <1> Completed Suicide: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - <1> Completed Suicide | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - <2> Suicide Attempt: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - <2> Suicide Attempt | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - <3> Preparatory Acts Towards Imminent Suicidal Behavior: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - <3> Preparatory Acts Towards Imminent Suicidal Behavior | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - <4> Suicidal Ideation: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - <4> Suicidal Ideation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - <7> Self-injurious Behavior, No Suicidal Intent: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - <7> Self-injurious Behavior, No Suicidal Intent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Response to Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 is a 9 item self-report scale for the assessment of depressive symptoms. The PHQ-9 were completed by participants and reviewed by site staff at the pre-defined time points.
Time Frame: Week 0, 2, 4, 6, 8, 10, 12, 13-14.
Population: Safety analysis set included all participants randomly assigned to study treatment and who took at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (T2DM) | Placebo (Non-diabetic Obesity) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Number analyzed (Participants) | 16 | 6 | 20 | 22 | 22 | 22 | 21 | 22
Participants
  Week 0 - Little Interest/Pleasure in Things - Not At All: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Little Interest/Pleasure in Things - Not At All | 15 | 6 | 16 | 20 | 20 | 20 | 19 | 21
  Week 0 - Little Interest/Pleasure in Things - Several Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Little Interest/Pleasure in Things - Several Days | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 1
  Week 0 - Little Interest/Pleasure in Things - More Than Half the Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Little Interest/Pleasure in Things - More Than Half the Days | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
  Week 0 - Little Interest/Pleasure in Things - Nearly Every Day: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Little Interest/Pleasure in Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - Feeling Down Depressed or Hopeless - Not At All: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Feeling Down Depressed or Hopeless - Not At All | 14 | 6 | 19 | 18 | 19 | 22 | 19 | 19
  Week 0 - Feeling Down Depressed or Hopeless - Several Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Feeling Down Depressed or Hopeless - Several Days | 2 | 0 | 1 | 3 | 1 | 0 | 2 | 3
  Week 0 - Feeling Down Depressed or Hopeless - More Than Half the Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Feeling Down Depressed or Hopeless - More Than Half the Days | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Week 0 - Feeling Down Depressed or Hopeless - Nearly Every Day: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Feeling Down Depressed or Hopeless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - Trouble Falling or Staying Asleep - Not At All: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Trouble Falling or Staying Asleep - Not At All | 15 | 5 | 13 | 16 | 17 | 17 | 17 | 15
  Week 0 - Trouble Falling or Staying Asleep - Several Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Trouble Falling or Staying Asleep - Several Days | 1 | 0 | 5 | 4 | 2 | 4 | 2 | 7
  Week 0 - Trouble Falling or Staying Asleep - More Than Half the Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Trouble Falling or Staying Asleep - More Than Half the Days | 0 | 1 | 2 | 1 | 2 | 1 | 1 | 0
  Week 0 - Trouble Falling or Staying Asleep - Nearly Every Day: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Trouble Falling or Staying Asleep - Nearly Every Day | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Week 0 - Feeling Tired or Little Energy - Not At All: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Feeling Tired or Little Energy - Not At All | 13 | 3 | 13 | 15 | 17 | 16 | 14 | 15
  Week 0 - Feeling Tired or Little Energy - Several Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Feeling Tired or Little Energy - Several Days | 3 | 2 | 5 | 4 | 4 | 4 | 6 | 7
  Week 0 - Feeling Tired or Little Energy - More Than Half the Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Feeling Tired or Little Energy - More Than Half the Days | 0 | 1 | 2 | 2 | 0 | 2 | 1 | 0
  Week 0 - Feeling Tired or Little Energy - Nearly Every Day: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Feeling Tired or Little Energy - Nearly Every Day | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Week 0 - Poor Appetite or Overeating - Not At All: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Poor Appetite or Overeating - Not At All | 15 | 3 | 13 | 19 | 18 | 19 | 21 | 20
  Week 0 - Poor Appetite or Overeating - Several Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Poor Appetite or Overeating - Several Days | 1 | 2 | 6 | 1 | 3 | 2 | 0 | 1
  Week 0 - Poor Appetite or Overeating - More Than Half the Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Poor Appetite or Overeating - More Than Half the Days | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1
  Week 0 - Poor Appetite or Overeating - Nearly Every Day: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Poor Appetite or Overeating - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - Feeling Bad About Yourself - Not At All: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Feeling Bad About Yourself - Not At All | 16 | 6 | 20 | 22 | 20 | 22 | 21 | 21
  Week 0 - Feeling Bad About Yourself - Several Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Feeling Bad About Yourself - Several Days | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Week 0 - Feeling Bad About Yourself - More Than Half the Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Feeling Bad About Yourself - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - Feeling Bad About Yourself - Nearly Every Day: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Feeling Bad About Yourself - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - Trouble Concentrating on Things - Not At All: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Trouble Concentrating on Things - Not At All | 16 | 5 | 16 | 21 | 19 | 20 | 21 | 20
  Week 0 - Trouble Concentrating on Things - Several Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Trouble Concentrating on Things - Several Days | 0 | 1 | 3 | 1 | 1 | 2 | 0 | 2
  Week 0 - Trouble Concentrating on Things - More Than Half the Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Trouble Concentrating on Things - More Than Half the Days | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Week 0 - Trouble Concentrating on Things - Nearly Every Day: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Trouble Concentrating on Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - Moving Slowly or Fidgety/Restless - Not At All: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Moving Slowly or Fidgety/Restless - Not At All | 16 | 6 | 19 | 22 | 21 | 21 | 21 | 21
  Week 0 - Moving Slowly or Fidgety/Restless - Several Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Moving Slowly or Fidgety/Restless - Several Days | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  Week 0 - Moving Slowly or Fidgety/Restless - More Than Half the Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Moving Slowly or Fidgety/Restless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - Moving Slowly or Fidgety/Restless - Nearly Every Day: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Moving Slowly or Fidgety/Restless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - Thoughts You Be Better Off Dead - Not At All: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Thoughts You Be Better Off Dead - Not At All | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Thoughts You Be Better Off Dead - Several Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Thoughts You Be Better Off Dead - Several Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - Thoughts You Be Better Off Dead - More Than Half the Days: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Thoughts You Be Better Off Dead - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 0 - Thoughts You Be Better Off Dead - Nearly Every Day: number analyzed (Participants) | 16 | 6 | 20 | 22 | 21 | 22 | 21 | 22
  Week 0 - Thoughts You Be Better Off Dead - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - Little Interest/Pleasure in Things - Not At All: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Little Interest/Pleasure in Things - Not At All | 13 | 5 | 16 | 17 | 21 | 19 | 16 | 18
  Week 2 - Little Interest/Pleasure in Things - Several Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Little Interest/Pleasure in Things - Several Days | 1 | 1 | 4 | 2 | 0 | 2 | 2 | 1
  Week 2 - Little Interest/Pleasure in Things - More Than Half the Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Little Interest/Pleasure in Things - More Than Half the Days | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Week 2 - Little Interest/Pleasure in Things - Nearly Every Day: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Little Interest/Pleasure in Things - Nearly Every Day | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Week 2 - Feeling Down Depressed or Hopeless - Not At All: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Feeling Down Depressed or Hopeless - Not At All | 12 | 6 | 18 | 20 | 21 | 21 | 17 | 18
  Week 2 - Feeling Down Depressed or Hopeless - Several Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Feeling Down Depressed or Hopeless - Several Days | 2 | 0 | 2 | 1 | 0 | 0 | 2 | 2
  Week 2 - Feeling Down Depressed or Hopeless - More Than Half the Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Feeling Down Depressed or Hopeless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - Feeling Down Depressed or Hopeless - Nearly Every Day: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Feeling Down Depressed or Hopeless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - Trouble Falling or Staying Asleep - Not At All: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Trouble Falling or Staying Asleep - Not At All | 14 | 4 | 14 | 16 | 19 | 17 | 13 | 15
  Week 2 - Trouble Falling or Staying Asleep - Several Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Trouble Falling or Staying Asleep - Several Days | 0 | 1 | 5 | 2 | 2 | 3 | 4 | 5
  Week 2 - Trouble Falling or Staying Asleep - More Than Half the Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Trouble Falling or Staying Asleep - More Than Half the Days | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
  Week 2 - Trouble Falling or Staying Asleep - Nearly Every Day: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Trouble Falling or Staying Asleep - Nearly Every Day | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
  Week 2 - Feeling Tired or Little Energy - Not At All: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Feeling Tired or Little Energy - Not At All | 11 | 3 | 13 | 17 | 18 | 17 | 16 | 14
  Week 2 - Feeling Tired or Little Energy - Several Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Feeling Tired or Little Energy - Several Days | 3 | 2 | 6 | 2 | 3 | 3 | 2 | 5
  Week 2 - Feeling Tired or Little Energy - More Than Half the Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Feeling Tired or Little Energy - More Than Half the Days | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1
  Week 2 - Feeling Tired or Little Energy - Nearly Every Day: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Feeling Tired or Little Energy - Nearly Every Day | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 2 - Poor Appetite or Overeating - Not At All: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Poor Appetite or Overeating - Not At All | 12 | 2 | 15 | 15 | 19 | 18 | 17 | 17
  Week 2 - Poor Appetite or Overeating - Several Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Poor Appetite or Overeating - Several Days | 2 | 3 | 4 | 6 | 2 | 2 | 2 | 2
  Week 2 - Poor Appetite or Overeating - More Than Half the Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Poor Appetite or Overeating - More Than Half the Days | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Week 2 - Poor Appetite or Overeating - Nearly Every Day: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Poor Appetite or Overeating - Nearly Every Day | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 2 - Feeling Bad About Yourself - Not At All: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Feeling Bad About Yourself - Not At All | 14 | 6 | 18 | 21 | 21 | 20 | 19 | 19
  Week 2 - Feeling Bad About Yourself - Several Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Feeling Bad About Yourself - Several Days | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  Week 2 - Feeling Bad About Yourself - More Than Half the Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Feeling Bad About Yourself - More Than Half the Days | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 2 - Feeling Bad About Yourself - Nearly Every Day: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Feeling Bad About Yourself - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - Trouble Concentrating on Things - Not At All: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Trouble Concentrating on Things - Not At All | 14 | 5 | 17 | 20 | 20 | 19 | 18 | 18
  Week 2 - Trouble Concentrating on Things - Several Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Trouble Concentrating on Things - Several Days | 0 | 0 | 2 | 1 | 1 | 2 | 1 | 2
  Week 2 - Trouble Concentrating on Things - More Than Half the Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Trouble Concentrating on Things - More Than Half the Days | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - Trouble Concentrating on Things - Nearly Every Day: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Trouble Concentrating on Things - Nearly Every Day | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 2 - Moving Slowly or Fidgety/Restless - Not At All: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Moving Slowly or Fidgety/Restless - Not At All | 14 | 5 | 19 | 20 | 21 | 21 | 18 | 20
  Week 2 - Moving Slowly or Fidgety/Restless - Several Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Moving Slowly or Fidgety/Restless - Several Days | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Week 2 - Moving Slowly or Fidgety/Restless - More Than Half the Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Moving Slowly or Fidgety/Restless - More Than Half the Days | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Week 2 - Moving Slowly or Fidgety/Restless - Nearly Every Day: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Moving Slowly or Fidgety/Restless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - Thoughts You Be Better Off Dead - Not At All: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Thoughts You Be Better Off Dead - Not At All | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Thoughts You Be Better Off Dead - Several Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Thoughts You Be Better Off Dead - Several Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - Thoughts You Be Better Off Dead - More Than Half the Days: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Thoughts You Be Better Off Dead - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 - Thoughts You Be Better Off Dead - Nearly Every Day: number analyzed (Participants) | 14 | 6 | 20 | 21 | 21 | 21 | 19 | 20
  Week 2 - Thoughts You Be Better Off Dead - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - Little Interest/Pleasure in Things - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Little Interest/Pleasure in Things - Not At All | 12 | 4 | 16 | 20 | 21 | 19 | 18 | 16
  Week 4 - Little Interest/Pleasure in Things - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Little Interest/Pleasure in Things - Several Days | 2 | 0 | 3 | 0 | 0 | 3 | 1 | 1
  Week 4 - Little Interest/Pleasure in Things - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Little Interest/Pleasure in Things - More Than Half the Days | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Week 4 - Little Interest/Pleasure in Things - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Little Interest/Pleasure in Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 -Feeling Down Depressed or Hopeless - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 -Feeling Down Depressed or Hopeless - Not At All | 13 | 5 | 18 | 18 | 21 | 22 | 18 | 15
  Week 4 - Feeling Down Depressed or Hopeless - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Feeling Down Depressed or Hopeless - Several Days | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 2
  Week 4 - Feeling Down Depressed or Hopeless - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Feeling Down Depressed or Hopeless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - Feeling Down Depressed or Hopeless - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Feeling Down Depressed or Hopeless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - Trouble Falling or Staying Asleep - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Trouble Falling or Staying Asleep - Not At All | 13 | 3 | 11 | 14 | 20 | 18 | 16 | 14
  Week 4 - Trouble Falling or Staying Asleep - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Trouble Falling or Staying Asleep - Several Days | 1 | 1 | 8 | 4 | 1 | 4 | 2 | 3
  Week 4 - Trouble Falling or Staying Asleep - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Trouble Falling or Staying Asleep - More Than Half the Days | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Week 4 - Trouble Falling or Staying Asleep - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Trouble Falling or Staying Asleep - Nearly Every Day | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Week 4 - Feeling Tired or Little Energy - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Feeling Tired or Little Energy - Not At All | 11 | 2 | 10 | 17 | 18 | 17 | 14 | 9
  Week 4 - Feeling Tired or Little Energy - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Feeling Tired or Little Energy - Several Days | 3 | 1 | 8 | 2 | 1 | 5 | 4 | 8
  Week 4 - Feeling Tired or Little Energy - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Feeling Tired or Little Energy - More Than Half the Days | 0 | 2 | 1 | 2 | 2 | 0 | 0 | 0
  Week 4 - Feeling Tired or Little Energy - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Feeling Tired or Little Energy - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 4 - Poor Appetite or Overeating - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Poor Appetite or Overeating - Not At All | 11 | 3 | 14 | 18 | 20 | 16 | 16 | 13
  Week 4 - Poor Appetite or Overeating - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Poor Appetite or Overeating - Several Days | 3 | 2 | 3 | 3 | 0 | 3 | 2 | 2
  Week 4 - Poor Appetite or Overeating - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Poor Appetite or Overeating - More Than Half the Days | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1
  Week 4 - Poor Appetite or Overeating - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Poor Appetite or Overeating - Nearly Every Day | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Week 4 - Feeling Bad About Yourself - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Feeling Bad About Yourself - Not At All | 14 | 5 | 19 | 21 | 21 | 22 | 18 | 17
  Week 4 - Feeling Bad About Yourself - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Feeling Bad About Yourself - Several Days | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 4 - Feeling Bad About Yourself - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Feeling Bad About Yourself - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - Feeling Bad About Yourself - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Feeling Bad About Yourself - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - Trouble Concentrating on Things - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Trouble Concentrating on Things - Not At All | 13 | 4 | 16 | 20 | 20 | 21 | 19 | 16
  Week 4 - Trouble Concentrating on Things - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Trouble Concentrating on Things - Several Days | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 1
  Week 4 - Trouble Concentrating on Things - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Trouble Concentrating on Things - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - Trouble Concentrating on Things - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Trouble Concentrating on Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - Moving Slowly or Fidgety/Restless - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Moving Slowly or Fidgety/Restless - Not At All | 14 | 4 | 18 | 20 | 21 | 21 | 19 | 17
  Week 4 - Moving Slowly or Fidgety/Restless - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Moving Slowly or Fidgety/Restless - Several Days | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
  Week 4 - Moving Slowly or Fidgety/Restless - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Moving Slowly or Fidgety/Restless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - Moving Slowly or Fidgety/Restless - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Moving Slowly or Fidgety/Restless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - Thoughts You Be Better Off Dead - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Thoughts You Be Better Off Dead - Not At All | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Thoughts You Be Better Off Dead - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Thoughts You Be Better Off Dead - Several Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - Thoughts You Be Better Off Dead - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Thoughts You Be Better Off Dead - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 - Thoughts You Be Better Off Dead - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 21 | 21 | 22 | 19 | 17
  Week 4 - Thoughts You Be Better Off Dead - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 -Little Interest/Pleasure in Things - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Little Interest/Pleasure in Things - Not At All | 12 | 4 | 15 | 17 | 19 | 16 | 14 | 14
  Week 6 -Little Interest/Pleasure in Things - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Little Interest/Pleasure in Things - Several Days | 2 | 1 | 4 | 2 | 0 | 3 | 1 | 1
  Week 6 -Little Interest/Pleasure in Things - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Little Interest/Pleasure in Things - More Than Half the Days | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Week 6 -Little Interest/Pleasure in Things - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Little Interest/Pleasure in Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 -Feeling Down Depressed or Hopeless - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Down Depressed or Hopeless - Not At All | 12 | 5 | 18 | 20 | 18 | 18 | 15 | 13
  Week 6 -Feeling Down Depressed or Hopeless - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Down Depressed or Hopeless - Several Days | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 2
  Week 6 -Feeling Down Depressed or Hopeless - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Down Depressed or Hopeless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 -Feeling Down Depressed or Hopeless - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Down Depressed or Hopeless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 -Trouble Falling or Staying Asleep - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Trouble Falling or Staying Asleep - Not At All | 12 | 4 | 12 | 14 | 16 | 18 | 12 | 10
  Week 6 -Trouble Falling or Staying Asleep - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Trouble Falling or Staying Asleep - Several Days | 1 | 0 | 7 | 6 | 3 | 1 | 3 | 4
  Week 6 -Trouble Falling or Staying Asleep - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Trouble Falling or Staying Asleep - More Than Half the Days | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Week 6 -Trouble Falling or Staying Asleep - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Trouble Falling or Staying Asleep - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 6 -Feeling Tired or Little Energy - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Tired or Little Energy - Not At All | 12 | 2 | 11 | 16 | 15 | 15 | 10 | 10
  Week 6 -Feeling Tired or Little Energy - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Tired or Little Energy - Several Days | 2 | 2 | 7 | 3 | 4 | 4 | 5 | 5
  Week 6 -Feeling Tired or Little Energy - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Tired or Little Energy - More Than Half the Days | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
  Week 6 -Feeling Tired or Little Energy - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Tired or Little Energy - Nearly Every Day | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 6 -Poor Appetite or Overeating - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Poor Appetite or Overeating - Not At All | 12 | 2 | 14 | 14 | 15 | 13 | 9 | 12
  Week 6 -Poor Appetite or Overeating - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Poor Appetite or Overeating - Several Days | 2 | 2 | 4 | 6 | 3 | 3 | 6 | 3
  Week 6 -Poor Appetite or Overeating - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Poor Appetite or Overeating - More Than Half the Days | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0
  Week 6 -Poor Appetite or Overeating - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Poor Appetite or Overeating - Nearly Every Day | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 6 -Feeling Bad About Yourself - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Bad About Yourself - Not At All | 14 | 5 | 18 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Bad About Yourself - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Bad About Yourself - Several Days | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 6 -Feeling Bad About Yourself - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Bad About Yourself - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 -Feeling Bad About Yourself - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Feeling Bad About Yourself - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 -Trouble Concentrating on Things - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Trouble Concentrating on Things - Not At All | 13 | 4 | 14 | 19 | 19 | 18 | 16 | 14
  Week 6 -Trouble Concentrating on Things - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Trouble Concentrating on Things - Several Days | 1 | 1 | 5 | 1 | 0 | 1 | 0 | 1
  Week 6 -Trouble Concentrating on Things - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Trouble Concentrating on Things - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 -Trouble Concentrating on Things - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Trouble Concentrating on Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 -Moving Slowly or Fidgety/Restless - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Moving Slowly or Fidgety/Restless - Not At All | 14 | 5 | 18 | 20 | 19 | 18 | 16 | 15
  Week 6 -Moving Slowly or Fidgety/Restless - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Moving Slowly or Fidgety/Restless - Several Days | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Week 6 -Moving Slowly or Fidgety/Restless - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Moving Slowly or Fidgety/Restless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 -Moving Slowly or Fidgety/Restless - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 -Moving Slowly or Fidgety/Restless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 - Thoughts You Be Better Off Dead - Not At All: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 - Thoughts You Be Better Off Dead - Not At All | 14 | 5 | 18 | 20 | 19 | 19 | 16 | 15
  Week 6 - Thoughts You Be Better Off Dead - Several Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 - Thoughts You Be Better Off Dead - Several Days | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 6 - Thoughts You Be Better Off Dead - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 - Thoughts You Be Better Off Dead - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6 - Thoughts You Be Better Off Dead - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 19 | 20 | 19 | 19 | 16 | 15
  Week 6 - Thoughts You Be Better Off Dead - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Little Interest/Pleasure in Things - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Little Interest/Pleasure in Things - Not At All | 13 | 5 | 16 | 16 | 18 | 17 | 15 | 13
  Week 8 - Little Interest/Pleasure in Things - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Little Interest/Pleasure in Things - Several Days | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 2
  Week 8 - Little Interest/Pleasure in Things - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Little Interest/Pleasure in Things - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Little Interest/Pleasure in Things - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Little Interest/Pleasure in Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Feeling Down Depressed or Hopeless - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Feeling Down Depressed or Hopeless - Not At All | 14 | 5 | 18 | 17 | 16 | 18 | 15 | 14
  Week 8 - Feeling Down Depressed or Hopeless - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Feeling Down Depressed or Hopeless - Several Days | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1
  Week 8 - Feeling Down Depressed or Hopeless - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Feeling Down Depressed or Hopeless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Feeling Down Depressed or Hopeless - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Feeling Down Depressed or Hopeless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Trouble Falling or Staying Asleep - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Trouble Falling or Staying Asleep - Not At All | 13 | 3 | 12 | 13 | 15 | 17 | 13 | 10
  Week 8 - Trouble Falling or Staying Asleep - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Trouble Falling or Staying Asleep - Several Days | 1 | 1 | 5 | 5 | 3 | 1 | 2 | 5
  Week 8 - Trouble Falling or Staying Asleep - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Trouble Falling or Staying Asleep - More Than Half the Days | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Week 8 - Trouble Falling or Staying Asleep - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Trouble Falling or Staying Asleep - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 8 - Feeling Tired or Little Energy - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Feeling Tired or Little Energy - Not At All | 11 | 3 | 13 | 16 | 16 | 16 | 9 | 10
  Week 8 - Feeling Tired or Little Energy - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Feeling Tired or Little Energy - Several Days | 3 | 2 | 4 | 1 | 2 | 2 | 6 | 4
  Week 8 - Feeling Tired or Little Energy - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Feeling Tired or Little Energy - More Than Half the Days | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
  Week 8 - Feeling Tired or Little Energy - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Feeling Tired or Little Energy - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Poor Appetite or Overeating - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Poor Appetite or Overeating - Not At All | 11 | 2 | 15 | 13 | 15 | 13 | 9 | 12
  Week 8 - Poor Appetite or Overeating - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Poor Appetite or Overeating - Several Days | 3 | 2 | 3 | 5 | 3 | 3 | 4 | 3
  Week 8 - Poor Appetite or Overeating - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Poor Appetite or Overeating - More Than Half the Days | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0
  Week 8 - Poor Appetite or Overeating - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Poor Appetite or Overeating - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 8 - Feeling Bad About Yourself - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Feeling Bad About Yourself - Not At All | 14 | 5 | 18 | 18 | 18 | 18 | 15 | 14
  Week 8 - Feeling Bad About Yourself - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Feeling Bad About Yourself - Several Days | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Week 8 - Feeling Bad About Yourself - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Feeling Bad About Yourself - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Feeling Bad About Yourself - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Feeling Bad About Yourself - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Trouble Concentrating on Things - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Trouble Concentrating on Things - Not At All | 13 | 4 | 14 | 16 | 18 | 17 | 15 | 14
  Week 8 - Trouble Concentrating on Things - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Trouble Concentrating on Things - Several Days | 1 | 1 | 3 | 2 | 0 | 1 | 1 | 1
  Week 8 - Trouble Concentrating on Things - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Trouble Concentrating on Things - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Trouble Concentrating on Things - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Trouble Concentrating on Things - Nearly Every Day | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 8 - Moving Slowly or Fidgety/Restless - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Moving Slowly or Fidgety/Restless - Not At All | 14 | 5 | 17 | 18 | 18 | 18 | 16 | 15
  Week 8 - Moving Slowly or Fidgety/Restless - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Moving Slowly or Fidgety/Restless - Several Days | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 8 - Moving Slowly or Fidgety/Restless - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Moving Slowly or Fidgety/Restless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Moving Slowly or Fidgety/Restless - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Moving Slowly or Fidgety/Restless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Thoughts You Be Better Off Dead - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Thoughts You Be Better Off Dead - Not At All | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Thoughts You Be Better Off Dead - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Thoughts You Be Better Off Dead - Several Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Thoughts You Be Better Off Dead - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Thoughts You Be Better Off Dead - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 - Thoughts You Be Better Off Dead - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 18 | 18 | 16 | 15
  Week 8 - Thoughts You Be Better Off Dead - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - Little Interest/Pleasure in Things - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Little Interest/Pleasure in Things - Not At All | 13 | 5 | 17 | 15 | 16 | 16 | 14 | 13
  Week 10 - Little Interest/Pleasure in Things - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Little Interest/Pleasure in Things - Several Days | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2
  Week 10 - Little Interest/Pleasure in Things - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Little Interest/Pleasure in Things - More Than Half the Days | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Week 10 - Little Interest/Pleasure in Things - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Little Interest/Pleasure in Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - Feeling Down Depressed or Hopeless - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Feeling Down Depressed or Hopeless - Not At All | 13 | 5 | 18 | 16 | 15 | 17 | 14 | 14
  Week 10 - Feeling Down Depressed or Hopeless - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Feeling Down Depressed or Hopeless - Several Days | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 1
  Week 10 - Feeling Down Depressed or Hopeless - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Feeling Down Depressed or Hopeless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - Feeling Down Depressed or Hopeless - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Feeling Down Depressed or Hopeless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - Trouble Falling or Staying Asleep - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Trouble Falling or Staying Asleep - Not At All | 13 | 3 | 13 | 14 | 14 | 15 | 12 | 10
  Week 10 - Trouble Falling or Staying Asleep - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Trouble Falling or Staying Asleep - Several Days | 1 | 1 | 5 | 3 | 2 | 1 | 2 | 5
  Week 10 - Trouble Falling or Staying Asleep - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Trouble Falling or Staying Asleep - More Than Half the Days | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Week 10 - Trouble Falling or Staying Asleep - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Trouble Falling or Staying Asleep - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 10 - Feeling Tired or Little Energy - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Feeling Tired or Little Energy - Not At All | 11 | 2 | 11 | 14 | 14 | 13 | 12 | 9
  Week 10 - Feeling Tired or Little Energy - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Feeling Tired or Little Energy - Several Days | 3 | 2 | 7 | 3 | 2 | 2 | 2 | 5
  Week 10 - Feeling Tired or Little Energy - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Feeling Tired or Little Energy - More Than Half the Days | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1
  Week 10 - Feeling Tired or Little Energy - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Feeling Tired or Little Energy - Nearly Every Day | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Week 10 - Poor Appetite or Overeating - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Poor Appetite or Overeating - Not At All | 10 | 2 | 15 | 16 | 14 | 11 | 10 | 12
  Week 10 - Poor Appetite or Overeating - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Poor Appetite or Overeating - Several Days | 4 | 3 | 3 | 2 | 1 | 5 | 2 | 3
  Week 10 - Poor Appetite or Overeating - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Poor Appetite or Overeating - More Than Half the Days | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
  Week 10 - Poor Appetite or Overeating - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Poor Appetite or Overeating - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 10 - Feeling Bad About Yourself - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Feeling Bad About Yourself - Not At All | 14 | 5 | 18 | 18 | 16 | 17 | 14 | 15
  Week 10 - Feeling Bad About Yourself - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Feeling Bad About Yourself - Several Days | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 10 - Feeling Bad About Yourself - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Feeling Bad About Yourself - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - Feeling Bad About Yourself - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Feeling Bad About Yourself - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - Trouble Concentrating on Things - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Trouble Concentrating on Things - Not At All | 13 | 5 | 17 | 17 | 16 | 16 | 15 | 15
  Week 10 - Trouble Concentrating on Things - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Trouble Concentrating on Things - Several Days | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
  Week 10 - Trouble Concentrating on Things - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Trouble Concentrating on Things - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - Trouble Concentrating on Things - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Trouble Concentrating on Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - Moving Slowly or Fidgety/Restless - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Moving Slowly or Fidgety/Restless - Not At All | 14 | 5 | 17 | 17 | 16 | 16 | 15 | 15
  Week 10 - Moving Slowly or Fidgety/Restless - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Moving Slowly or Fidgety/Restless - Several Days | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Week 10 - Moving Slowly or Fidgety/Restless - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Moving Slowly or Fidgety/Restless - More Than Half the Days | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Week 10 - Moving Slowly or Fidgety/Restless - Nearly Every Day: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Moving Slowly or Fidgety/Restless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - Thoughts You Be Better Off Dead - Not At All: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Thoughts You Be Better Off Dead - Not At All | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Thoughts You Be Better Off Dead - Several Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Thoughts You Be Better Off Dead - Several Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - Thoughts You Be Better Off Dead - More Than Half the Days: number analyzed (Participants) | 14 | 5 | 18 | 18 | 16 | 17 | 15 | 15
  Week 10 - Thoughts You Be Better Off Dead - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10 - Thoughts You Be Better Off Dead - Nearly Every Day: number analyzed (Participants) | 16 | 6 | 20 | 22 | 22 | 22 | 15 | 15
  Week 10 - Thoughts You Be Better Off Dead - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Little Interest/Pleasure in Things - Not At All: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Little Interest/Pleasure in Things - Not At All | 11 | 5 | 15 | 14 | 16 | 16 | 13 | 14
  Week 12 - Little Interest/Pleasure in Things - Several Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Little Interest/Pleasure in Things - Several Days | 2 | 0 | 3 | 2 | 0 | 0 | 1 | 0
  Week 12 - Little Interest/Pleasure in Things - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Little Interest/Pleasure in Things - More Than Half the Days | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Week 12 - Little Interest/Pleasure in Things - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Little Interest/Pleasure in Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Feeling Down Depressed or Hopeless - Not At All: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Feeling Down Depressed or Hopeless - Not At All | 11 | 5 | 18 | 17 | 16 | 16 | 13 | 14
  Week 12 - Feeling Down Depressed or Hopeless - Several Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Feeling Down Depressed or Hopeless - Several Days | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Week 12 - Feeling Down Depressed or Hopeless - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Feeling Down Depressed or Hopeless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Feeling Down Depressed or Hopeless - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Feeling Down Depressed or Hopeless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Trouble Falling or Staying Asleep - Not At All: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Trouble Falling or Staying Asleep - Not At All | 11 | 3 | 12 | 12 | 15 | 14 | 12 | 9
  Week 12 - Trouble Falling or Staying Asleep - Several Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Trouble Falling or Staying Asleep - Several Days | 2 | 2 | 6 | 5 | 1 | 1 | 1 | 4
  Week 12 - Trouble Falling or Staying Asleep - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Trouble Falling or Staying Asleep - More Than Half the Days | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
  Week 12 - Trouble Falling or Staying Asleep - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Trouble Falling or Staying Asleep - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 12 - Feeling Tired or Little Energy - Not At All: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Feeling Tired or Little Energy - Not At All | 10 | 3 | 12 | 14 | 14 | 14 | 11 | 9
  Week 12 - Feeling Tired or Little Energy - Several Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Feeling Tired or Little Energy - Several Days | 3 | 2 | 6 | 3 | 2 | 2 | 3 | 5
  Week 12 - Feeling Tired or Little Energy - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Feeling Tired or Little Energy - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Feeling Tired or Little Energy - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Feeling Tired or Little Energy - Nearly Every Day | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Week 12 - Poor Appetite or Overeating - Not At All: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Poor Appetite or Overeating - Not At All | 10 | 2 | 14 | 13 | 14 | 14 | 9 | 12
  Week 12 - Poor Appetite or Overeating - Several Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Poor Appetite or Overeating - Several Days | 3 | 3 | 3 | 5 | 2 | 2 | 4 | 1
  Week 12 - Poor Appetite or Overeating - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Poor Appetite or Overeating - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Poor Appetite or Overeating - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Poor Appetite or Overeating - Nearly Every Day | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  Week 12 - Feeling Bad About Yourself - Not At All: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Feeling Bad About Yourself - Not At All | 13 | 5 | 18 | 18 | 16 | 16 | 13 | 14
  Week 12 - Feeling Bad About Yourself - Several Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Feeling Bad About Yourself - Several Days | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 12 - Feeling Bad About Yourself - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Feeling Bad About Yourself - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Feeling Bad About Yourself - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Feeling Bad About Yourself - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Trouble Concentrating on Things - Not At All: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Trouble Concentrating on Things - Not At All | 11 | 5 | 17 | 17 | 16 | 16 | 14 | 14
  Week 12 - Trouble Concentrating on Things - Several Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Trouble Concentrating on Things - Several Days | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 12 - Trouble Concentrating on Things - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Trouble Concentrating on Things - More Than Half the Days | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Week 12 - Trouble Concentrating on Things - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Trouble Concentrating on Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Moving Slowly or Fidgety/Restless - Not At All: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Moving Slowly or Fidgety/Restless - Not At All | 12 | 5 | 17 | 18 | 16 | 16 | 14 | 14
  Week 12 - Moving Slowly or Fidgety/Restless - Several Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Moving Slowly or Fidgety/Restless - Several Days | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 12 - Moving Slowly or Fidgety/Restless - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Moving Slowly or Fidgety/Restless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Moving Slowly or Fidgety/Restless - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Moving Slowly or Fidgety/Restless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Thoughts You Be Better Off Dead - Not At All: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Thoughts You Be Better Off Dead - Not At All | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Thoughts You Be Better Off Dead - Several Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Thoughts You Be Better Off Dead - Several Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Thoughts You Be Better Off Dead - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Thoughts You Be Better Off Dead - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12 - Thoughts You Be Better Off Dead - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 18 | 18 | 16 | 16 | 14 | 14
  Week 12 - Thoughts You Be Better Off Dead - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Little Interest/Pleasure in Things - Not At All: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Little Interest/Pleasure in Things - Not At All | 11 | 5 | 14 | 17 | 16 | 17 | 13 | 12
  Follow-Up - Little Interest/Pleasure in Things - Several Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Little Interest/Pleasure in Things - Several Days | 2 | 0 | 3 | 1 | 0 | 0 | 1 | 1
  Follow-Up - Little Interest/Pleasure in Things - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Little Interest/Pleasure in Things - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Follow-Up - Little Interest/Pleasure in Things - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Little Interest/Pleasure in Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Feeling Down Depressed or Hopeless - Not At All: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Feeling Down Depressed or Hopeless - Not At All | 13 | 5 | 17 | 17 | 16 | 16 | 13 | 12
  Follow-Up - Feeling Down Depressed or Hopeless - Several Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Feeling Down Depressed or Hopeless - Several Days | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
  Follow-Up - Feeling Down Depressed or Hopeless - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Feeling Down Depressed or Hopeless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Feeling Down Depressed or Hopeless - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Feeling Down Depressed or Hopeless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Trouble Falling or Staying Asleep - Not At All: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Trouble Falling or Staying Asleep - Not At All | 12 | 4 | 12 | 13 | 14 | 15 | 12 | 9
  Follow-Up - Trouble Falling or Staying Asleep - Several Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Trouble Falling or Staying Asleep - Several Days | 0 | 1 | 5 | 5 | 2 | 2 | 1 | 4
  Follow-Up - Trouble Falling or Staying Asleep - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Trouble Falling or Staying Asleep - More Than Half the Days | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Trouble Falling or Staying Asleep - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Trouble Falling or Staying Asleep - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Follow-Up - Feeling Tired or Little Energy - Not At All: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Feeling Tired or Little Energy - Not At All | 11 | 2 | 11 | 14 | 14 | 17 | 12 | 9
  Follow-Up - Feeling Tired or Little Energy - Several Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Feeling Tired or Little Energy - Several Days | 2 | 3 | 5 | 4 | 2 | 0 | 2 | 4
  Follow-Up - Feeling Tired or Little Energy - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Feeling Tired or Little Energy - More Than Half the Days | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Follow-Up - Feeling Tired or Little Energy - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Feeling Tired or Little Energy - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Poor Appetite or Overeating - Not At All: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Poor Appetite or Overeating - Not At All | 11 | 3 | 13 | 16 | 15 | 16 | 12 | 12
  Follow-Up - Poor Appetite or Overeating - Several Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Poor Appetite or Overeating - Several Days | 2 | 2 | 4 | 2 | 1 | 1 | 2 | 1
  Follow-Up - Poor Appetite or Overeating - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Poor Appetite or Overeating - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Follow-Up - Poor Appetite or Overeating - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Poor Appetite or Overeating - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Feeling Bad About Yourself - Not At All: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Feeling Bad About Yourself - Not At All | 13 | 5 | 17 | 18 | 16 | 17 | 13 | 13
  Follow-Up - Feeling Bad About Yourself - Several Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Feeling Bad About Yourself - Several Days | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Follow-Up - Feeling Bad About Yourself - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Feeling Bad About Yourself - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Follow-Up - Feeling Bad About Yourself - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Feeling Bad About Yourself - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Trouble Concentrating on Things - Not At All: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Trouble Concentrating on Things - Not At All | 12 | 5 | 17 | 16 | 16 | 17 | 14 | 13
  Follow-Up - Trouble Concentrating on Things - Several Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Trouble Concentrating on Things - Several Days | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
  Follow-Up - Trouble Concentrating on Things - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Trouble Concentrating on Things - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Trouble Concentrating on Things - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Trouble Concentrating on Things - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Moving Slowly or Fidgety/Restless - Not At All: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Moving Slowly or Fidgety/Restless - Not At All | 12 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Moving Slowly or Fidgety/Restless - Several Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Moving Slowly or Fidgety/Restless - Several Days | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Moving Slowly or Fidgety/Restless - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Moving Slowly or Fidgety/Restless - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Moving Slowly or Fidgety/Restless - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Moving Slowly or Fidgety/Restless - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Thoughts You Be Better Off Dead - Not At All: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Thoughts You Be Better Off Dead - Not At All | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Thoughts You Be Better Off Dead - Several Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Thoughts You Be Better Off Dead - Several Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Thoughts You Be Better Off Dead - More Than Half the Days: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Thoughts You Be Better Off Dead - More Than Half the Days | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Follow-Up - Thoughts You Be Better Off Dead - Nearly Every Day: number analyzed (Participants) | 13 | 5 | 17 | 18 | 16 | 17 | 14 | 14
  Follow-Up - Thoughts You Be Better Off Dead - Nearly Every Day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline (CFB) in Fasting Plasma Glucose at Week 2
Description: Baseline was defined as the result closest prior to dosing at Day1. The MMRM model included treatment, time, strata (male versus female) and treatment-by-time interaction as fixed effects, baseline as a covariate and the baseline-by-time interaction with time fitted as a repeated effect and participant as a random effect. An unstructured covariance matrix was used to estimate the variances and covariance within participant across time points.
Time Frame: Baseline, Week 2
Population: Estimand Set 1A that all evaluable participants with T2DM randomly assigned to IP and who took at least 1 dose of IP. For participants who discontinued IP and/or received glycemic rescue medication, all subsequent values were censored.
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21
mg/dL | -5.63 [-19.00 to 7.74] | -3.32 [-14.62 to 7.97] | -23.04 [-34.05 to -12.03] | -36.48 [-47.44 to -25.52] | -39.29 [-50.23 to -28.35] | -25.15 [-36.59 to -13.72]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.5863, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = 2.31, 90% CI 2-sided [-15.23 to 19.85] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.0494, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -17.41, 90% CI 2-sided [-34.75 to -0.06] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0019, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -30.85, 90% CI 2-sided [-48.09 to -13.61] — Test = PF06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0009, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -33.66, 90% CI 2-sided [-51.00 to -16.32] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.0343, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -19.52, 90% CI 2-sided [-37.12 to -1.92] — Test = PF-06882961 Reference = Placebo

8. Secondary Outcome: CFB in Fasting Plasma Glucose at Week 4
Description: as for outcome 7
Time Frame: Baseline, Week 4
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21
mg/dL | -13.12 [-26.88 to 0.64] | -16.45 [-28.11 to -4.79] | -32.77 [-43.98 to -21.55] | -45.92 [-57.20 to -34.64] | -48.97 [-60.52 to -37.42] | -41.60 [-53.38 to -29.83]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.3804, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -3.33, 90% CI 2-sided [-21.41 to 14.76] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.0348, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -19.65, 90% CI 2-sided [-37.44 to -1.87] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0014, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -32.80, 90% CI 2-sided [-50.54 to -15.05] — Test = PF06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0007, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -35.85, 90% CI 2-sided [-53.90 to -17.81] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.0052, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -28.49, 90% CI 2-sided [-46.60 to -10.37] — Test = PF-06882961 Reference = Placebo

9. Secondary Outcome: CFB in Fasting Plasma Glucose at Week 6
Description: as for outcome 7
Time Frame: Baseline, Week 6
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21
mg/dL | -3.75 [-19.85 to 12.35] | -29.33 [-43.35 to -15.31] | -36.70 [-50.13 to -23.27] | -43.82 [-57.90 to -29.75] | -49.22 [-63.14 to -35.31] | -37.38 [-51.77 to -22.99]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.0250, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -25.58, 90% CI 2-sided [-46.97 to -4.18] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.0053, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -32.95, 90% CI 2-sided [-53.95 to -11.95] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0012, Mixed Models Analysis; MMRM; Mean Difference (Final Values) = -40.07, 90% CI 2-sided [-61.41 to -18.73] — Test = PF06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0003, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -45.47, 90% CI 2-sided [-66.85 to -24.10] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.0055, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -33.63, 90% CI 2-sided [-55.19 to -12.08] — Test = PF-06882961 Reference = Placebo

10. Secondary Outcome: CFB in Fasting Plasma Glucose at Week 8
Description: as for outcome 7
Time Frame: Baseline, Week 8
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21
mg/dL | -5.90 [-20.83 to 9.04] | -33.69 [-47.42 to -19.96] | -31.57 [-44.56 to -18.58] | -52.84 [-66.55 to -39.13] | -39.69 [-53.63 to -25.75] | -48.02 [-62.47 to -33.57]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.0127, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -27.79, 90% CI 2-sided [-48.12 to -7.47] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.0171, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -25.67, 90% CI 2-sided [-45.51 to -5.83] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0001, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -46.94, 90% CI 2-sided [-67.16 to -26.72] — Test = PF06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0037, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -33.79, 90% CI 2-sided [-54.32 to -13.27] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.0005, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -42.13, 90% CI 2-sided [-62.85 to -21.40] — Test = PF-06882961 Reference = Placebo

11. Secondary Outcome: CFB in Fasting Plasma Glucose at Week 10
Description: as for outcome 7
Time Frame: Baseline, Week 10
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21
mg/dL | -23.39 [-39.07 to -7.71] | -36.24 [-51.69 to -20.78] | -38.21 [-52.17 to -24.26] | -57.36 [-72.43 to -42.29] | -22.08 [-36.88 to -7.29] | -37.81 [-53.52 to -22.11]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.1678, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -12.85, 90% CI 2-sided [-34.90 to 9.21] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.1223, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -14.82, 90% CI 2-sided [-35.85 to 6.21] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0054, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -33.97, 90% CI 2-sided [-55.66 to -12.28] — Test = PF06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.5398, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = 1.31, 90% CI 2-sided [-20.38 to 22.99] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.1409, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -14.42, 90% CI 2-sided [-36.56 to 7.72] — Test = PF-06882961 Reference = Placebo

12. Secondary Outcome: CFB in Fasting Plasma Glucose at Week 12
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21
mg/dL | -13.09 [-29.75 to 3.57] | -41.74 [-58.49 to -25.00] | -40.41 [-55.25 to -25.57] | -53.94 [-70.26 to -37.63] | -23.34 [-39.52 to -7.17] | -37.48 [-55.27 to -19.69]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.0236, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -28.65, 90% CI 2-sided [-52.31 to -4.99] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.0226, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -27.32, 90% CI 2-sided [-49.67 to -4.97] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0022, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -40.85, 90% CI 2-sided [-64.11 to -17.59] — Test = PF06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.2335, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -10.25, 90% CI 2-sided [-33.59 to 13.08] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.0494, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -24.38, 90% CI 2-sided [-48.69 to -0.08] — Test = PF-06882961 Reference = Placebo

13. Secondary Outcome: CFB in Glycolated Hemoglobin A1c (HbA1c) at Week 2
Description: as for outcome 7
Time Frame: Baseline, Week 2
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21
Percentage | -0.03 [-0.20 to 0.14] | -0.12 [-0.26 to 0.02] | -0.29 [-0.43 to -0.15] | -0.37 [-0.51 to -0.24] | -0.35 [-0.49 to -0.21] | -0.20 [-0.34 to -0.05]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.2485, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.09, 90% CI 2-sided [-0.31 to 0.13] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.0252, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.26, 90% CI 2-sided [-0.48 to -0.04] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0053, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.34, 90% CI 2-sided [-0.56 to -0.12] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0090, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.32, 90% CI 2-sided [-0.54 to -0.10] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.1066, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.17, 90% CI 2-sided [-0.39 to 0.05] — Test = PF-06882961 Reference = Placebo

14. Secondary Outcome: CFB in Glycolated HbA1c at Week 4
Description: as for outcome 7
Time Frame: Baseline, Week 4
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21
Percentage | -0.22 [-0.45 to 0.00] | -0.33 [-0.52 to -0.14] | -0.59 [-0.77 to -0.41] | -0.81 [-1.00 to -0.63] | -0.75 [-0.94 to -0.56] | -0.58 [-0.78 to -0.39]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.2740, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.11, 90% CI 2-sided [-0.40 to 0.19] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.0196, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.37, 90% CI 2-sided [-0.66 to -0.08] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0006, Mixed Models Analysis; MMRM; Mean Difference (Final Values) = -0.59, 90% CI 2-sided [-0.88 to -0.30] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0019, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.53, 90% CI 2-sided [-0.82 to -0.23] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.0243, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.36, 90% CI 2-sided [-0.66 to -0.06] — Test = PF-06882961 Reference = Placebo

15. Secondary Outcome: CFB in Glycolated HbA1c at Week 6
Description: as for outcome 7
Time Frame: Baseline, Week 6
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21
Percentage | -0.26 [-0.56 to 0.04] | -0.49 [-0.75 to -0.24] | -0.92 [-1.16 to -0.67] | -1.11 [-1.36 to -0.86] | -0.97 [-1.22 to -0.72] | -0.93 [-1.19 to -0.68]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.1587, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.23, 90% CI 2-sided [-0.62 to 0.15] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.0027, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.66, 90% CI 2-sided [-1.04 to -0.27] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0002, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.85, 90% CI 2-sided [-1.24 to -0.47] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0016, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.71, 90% CI 2-sided [-1.10 to -0.32] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.0027, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.67, 90% CI 2-sided [-1.07 to -0.28] — Test = PF-06882961 Reference = Placebo

16. Secondary Outcome: CFB in Glycolated HbA1c at Week 8
Description: as for outcome 7
Time Frame: Baseline, Week 8
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21
Percentage | -0.27 [-0.60 to 0.05] | -0.71 [-0.99 to -0.43] | -1.14 [-1.41 to -0.88] | -1.38 [-1.65 to -1.10] | -1.20 [-1.48 to -0.92] | -1.18 [-1.47 to -0.89]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.0472, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.43, 90% CI 2-sided [-0.86 to -0.01] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.0004, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.87, 90% CI 2-sided [-1.29 to -0.45] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p < 0.0001, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -1.10, 90% CI 2-sided [-1.53 to -0.68] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0003, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.93, 90% CI 2-sided [-1.36 to -0.50] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.0004, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.91, 90% CI 2-sided [-1.34 to -0.47] — Test = PF-06882961 Reference = Placebo

17. Secondary Outcome: CFB in Glycolated HbA1c at Week 10
Description: as for outcome 7
Time Frame: Baseline, Week 10
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21
Percentage | -0.32 [-0.69 to 0.05] | -1.00 [-1.33 to -0.67] | -1.26 [-1.57 to -0.95] | -1.48 [-1.81 to -1.16] | -1.22 [-1.55 to -0.89] | -1.36 [-1.70 to -1.03]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.0116, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.69, 90% CI 2-sided [-1.18 to -0.19] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.0008, Mixed Models Analysis; MMRM; Mean Difference (Final Values) = -0.94, 90% CI 2-sided [-1.43 to -0.46] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p < 0.0001, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -1.16, 90% CI 2-sided [-1.66 to -0.67] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0017, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.90, 90% CI 2-sided [-1.40 to -0.40] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.0004, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -1.05, 90% CI 2-sided [-1.55 to -0.55] — Test = PF-06882961 Reference = Placebo

18. Secondary Outcome: CFB in Glycolated HbA1c at Week 12
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 16 | 20 | 22 | 22 | 22 | 21
Percentage | -0.32 [-0.73 to 0.10] | -1.07 [-1.45 to -0.70] | -1.32 [-1.67 to -0.97] | -1.56 [-1.94 to -1.19] | -1.04 [-1.42 to -0.67] | -1.57 [-1.96 to -1.18]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.0132, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.76, 90% CI 2-sided [-1.32 to -0.20] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.0014, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -1.00, 90% CI 2-sided [-1.55 to -0.46] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0002, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -1.25, 90% CI 2-sided [-1.80 to -0.69] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0174, Mixed Models Analysis; MMRM; Mean Difference (Final Values) = -0.73, 90% CI 2-sided [-1.29 to -0.16] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.0002, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -1.25, 90% CI 2-sided [-1.82 to -0.69] — Test = PF-06882961 Reference = Placebo

19. Secondary Outcome: CFB in Body Weight at Week 2 (Participants With T2DM)
Description: Baseline was defined as the average of a duplicate measurement closest prior to dosing at Day 1. The MMRM model included treatment, time, strata (male versus female) and treatment-by-time interaction as fixed effects, baseline as a covariate and the baseline-by-time interaction with time fitted as a repeated effect and participant as a random effect. An unstructured covariance matrix was used to estimate the variances and covariance within participant across time points. Average of the duplicate measurements (where applicable) was used in analyses.
Time Frame: Baseline, Week 2
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 20 | 22 | 22 | 22 | 22 | 21
kg | -0.14 [-0.72 to 0.44] | -0.40 [-0.89 to 0.08] | -0.22 [-0.70 to 0.26] | -0.46 [-0.94 to 0.02] | -0.63 [-1.11 to -0.16] | -0.21 [-0.72 to 0.30]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.2843, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.26, 90% CI 2-sided [-1.02 to 0.50] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.4310, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.08, 90% CI 2-sided [-0.84 to 0.68] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.2402, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.32, 90% CI 2-sided [-1.07 to 0.43] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.1397, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.49, 90% CI 2-sided [-1.24 to 0.26] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.4393, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.07, 90% CI 2-sided [-0.85 to 0.71] — Test = PF-06882961 Reference = Placebo

20. Secondary Outcome: CFB in Body Weight at Week 4 (Participants With T2DM)
Description: as for outcome 19
Time Frame: Baseline, Week 4
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 20 | 22 | 22 | 22 | 22 | 21
kg | -0.46 [-1.40 to 0.47] | -1.23 [-2.03 to -0.44] | -0.34 [-1.11 to 0.43] | -1.58 [-2.35 to -0.81] | -1.47 [-2.25 to -0.70] | -0.41 [-1.23 to 0.41]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.1491, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.77, 90% CI 2-sided [-2.00 to 0.45] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.5664, Mixed Models Analysis — 1-Sided; MMRM; Median Difference (Final Values) = 0.12, 90% CI 2-sided [-1.09 to 1.34] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0632, Mixed Models Analysis — 1-Sided; MMRM; Median Difference (Final Values) = -1.12, 90% CI 2-sided [-2.33 to 0.09] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0847, Mixed Models Analysis — 1-Sided; MMRM; Median Difference (Final Values) = -1.01, 90% CI 2-sided [-2.23 to 0.20] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.5264, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = 0.05, 90% CI 2-sided [-1.20 to 1.30] — Test = PF-06882961 Reference = Placebo

21. Secondary Outcome: CFB in Body Weight at Week 6 (Participants With T2DM)
Description: as for outcome 19
Time Frame: Baseline, Week 6
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 20 | 22 | 22 | 22 | 22 | 21
kg | -0.38 [-1.42 to 0.66] | -1.86 [-2.77 to -0.95] | -0.65 [-1.52 to 0.23] | -2.74 [-3.65 to -1.83] | -2.23 [-3.13 to -1.33] | -1.16 [-2.10 to -0.21]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.0395, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -1.48, 90% CI 2-sided [-2.86 to -0.10] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.3726, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.27, 90% CI 2-sided [-1.63 to 1.10] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0028, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -2.36, 90% CI 2-sided [-3.74 to -0.98] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0139, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -1.85, 90% CI 2-sided [-3.23 to -0.47] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.1815, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.78, 90% CI 2-sided [-2.19 to 0.64] — Test = PF-06882961 Reference = Placebo

22. Secondary Outcome: CFB in Body Weight at Week 8 (Participants With T2DM)
Description: as for outcome 19
Time Frame: Baseline, Week 8
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 20 | 22 | 22 | 22 | 22 | 21
kg | -0.36 [-1.51 to 0.80] | -2.52 [-3.55 to -1.48] | -1.08 [-2.07 to -0.09] | -3.82 [-4.86 to -2.79] | -2.41 [-3.43 to -1.38] | -3.32 [-4.42 to -2.23]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.0112, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -2.16, 90% CI 2-sided [-3.71 to -0.61] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.2161, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.72, 90% CI 2-sided [-2.24 to 0.80] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p = 0.0002, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -3.47, 90% CI 2-sided [-5.02 to -1.92] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0147, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -2.05, 90% CI 2-sided [-3.59 to -0.51] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.0013, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -2.97, 90% CI 2-sided [-4.56 to -1.37] — Test = PF-06882961 Reference = Placebo

23. Secondary Outcome: CFB in Body Weight at Week 10 (Participants With T2DM)
Description: as for outcome 19
Time Frame: Baseline, Week 10
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 20 | 22 | 22 | 22 | 22 | 21
kg | -0.67 [-1.96 to 0.61] | -3.14 [-4.34 to -1.93] | -1.71 [-2.83 to -0.58] | -4.95 [-6.15 to -3.75] | -3.35 [-4.53 to -2.18] | -4.38 [-5.64 to -3.12]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.0111, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -2.46, 90% CI 2-sided [-4.22 to -0.70] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.1600, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -1.03, 90% CI 2-sided [-2.75 to 0.68] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p < 0.0001, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -4.27, 90% CI 2-sided [-6.03 to -2.52] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0061, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -2.68, 90% CI 2-sided [-4.42 to -0.94] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p = 0.0005, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -3.71, 90% CI 2-sided [-5.52 to -1.89] — Test = PF-06882961 Reference = Placebo

24. Secondary Outcome: CFB in Body Weight at Week 12 (Participants With T2DM)
Description: as for outcome 19
Time Frame: Baseline, Week 12
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo (T2DM) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM)
Number analyzed (Participants) | 20 | 22 | 22 | 22 | 22 | 21
kg | -0.42 [-1.87 to 1.03] | -3.64 [-5.03 to -2.24] | -1.93 [-3.22 to -0.64] | -5.38 [-6.77 to -3.98] | -2.93 [-4.29 to -1.56] | -5.37 [-6.86 to -3.88]
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID Low, Slow (T2DM); Test type: Superiority; p = 0.0047, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -3.21, 90% CI 2-sided [-5.22 to -1.20] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-06882961 80 mg BID High, Slow (T2DM); Test type: Superiority; p = 0.1003, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -1.51, 90% CI 2-sided [-3.45 to 0.44] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID Low, Fast (T2DM); Test type: Superiority; p < 0.0001, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -4.95, 90% CI 2-sided [-6.96 to -2.95] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-06882961 120 mg BID High, Fast (T2DM); Test type: Superiority; p = 0.0197, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -2.50, 90% CI 2-sided [-4.49 to -0.51] — Test = PF-06882961 Reference = Placebo
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-06882961 200 mg BID (T2DM); Test type: Superiority; p < 0.0001, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -4.94, 90% CI 2-sided [-7.03 to -2.85] — Test = PF-06882961 Reference = Placebo

25. Secondary Outcome: CFB in Body Weight at Week 2 (Non-diabetic Participants With Obesity)
Description: Body weight were measured in duplicate as indicated. The second weight measurement were obtained at least 1-2 minutes apart from the first weight measurement. Weight were recorded using a calibrated scale (with the same scale used if possible for the duration of the study) reporting weight in kilograms (kg), and accuracy to the nearest 0.1 kg; ie, the device distinguished a difference between 68.4 kg vs 68.3 kg. The scale was placed on a stable, flat surface. Weight measurement was taken under the following conditions: participant is in a fasted state; after void of urine; after removal of shoes, bulky layers of clothing and jackets so that only light clothing remained; while remaining was during the measurement.
Time Frame: Baseline, Week 2
Population: Estimand set 1B that all evaluable non-diabetic participants with obesity randomly assigned to IP and who took at least 1 dose of IP. For participants who discontinued IP, all subsequent values were censored.
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo (Non-diabetic Obesity) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Number analyzed (Participants) | 6 | 22
kg | 0.23 [-0.81 to 1.26] | -0.73 [-1.34 to -0.13]
Statistical Analysis 1: Comparison: Placebo (Non-diabetic Obesity) vs PF-06882961 200 mg BID (Non-diabetic Obesity); Test type: Superiority; p = 0.0836, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -0.96, 90% CI 2-sided [-2.12 to 0.19] — Test = PF-06882961 Reference = Placebo

26. Secondary Outcome: CFB in Body Weight at Week 4 (Non-diabetic Participants With Obesity)
Description: as for outcome 25
Time Frame: Baseline, Week 4
Population: as for outcome 25
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo (Non-diabetic Obesity) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Number analyzed (Participants) | 6 | 22
kg | 0.09 [-1.21 to 1.40] | -1.50 [-2.25 to -0.74]
Statistical Analysis 1: Comparison: Placebo (Non-diabetic Obesity) vs PF-06882961 200 mg BID (Non-diabetic Obesity); Test type: Superiority; p = 0.0386, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -1.59, 90% CI 2-sided [-3.07 to -0.12] — Test = PF-06882961 Reference = Placebo

27. Secondary Outcome: CFB in Body Weight at Week 6 (Non-diabetic Participants With Obesity)
Description: as for outcome 25
Time Frame: Baseline, Week 6
Population: as for outcome 25
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo (Non-diabetic Obesity) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Number analyzed (Participants) | 6 | 22
kg | -0.10 [-2.28 to 2.08] | -1.59 [-2.86 to -0.33]
Statistical Analysis 1: Comparison: Placebo (Non-diabetic Obesity) vs PF-06882961 200 mg BID (Non-diabetic Obesity); Test type: Superiority; p = 0.1566, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -1.50, 90% CI 2-sided [-3.99 to 1.00] — Test = PF-06882961 Reference = Placebo

28. Secondary Outcome: CFB in Body Weight at Week 8 (Non-diabetic Participants With Obesity)
Description: as for outcome 25
Time Frame: Baseline, Week 8
Population: as for outcome 25
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo (Non-diabetic Obesity) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Number analyzed (Participants) | 6 | 22
kg | 0.26 [-2.57 to 3.09] | -2.36 [-4.08 to -0.65]
Statistical Analysis 1: Comparison: Placebo (Non-diabetic Obesity) vs PF-06882961 200 mg BID (Non-diabetic Obesity); Test type: Superiority; p = 0.0916, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -2.62, 90% CI 2-sided [-5.91 to 0.67] — Test = PF-06882961 Reference = Placebo

29. Secondary Outcome: CFB in Body Weight at Week 10 (Non-diabetic Participants With Obesity)
Description: as for outcome 25
Time Frame: Baseline, Week 10
Population: as for outcome 25
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo (Non-diabetic Obesity) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Number analyzed (Participants) | 6 | 22
kg | -0.40 [-3.17 to 2.37] | -3.47 [-5.21 to -1.73]
Statistical Analysis 1: Comparison: Placebo (Non-diabetic Obesity) vs PF-06882961 200 mg BID (Non-diabetic Obesity); Test type: Superiority; p = 0.0590, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -3.07, 90% CI 2-sided [-6.31 to 0.17] — Test = PF-06882961 Reference = Placebo

30. Secondary Outcome: CFB in Body Weight at Week 12 (Non-diabetic Participants With Obesity)
Description: as for outcome 25
Time Frame: Baseline, Week 12
Population: as for outcome 25
Measure: Least Squares Mean (90% Confidence Interval); unit: kg
Arm/Group | Placebo (Non-diabetic Obesity) | PF-06882961 200 mg BID (Non-diabetic Obesity)
Number analyzed (Participants) | 6 | 22
kg | -0.11 [-3.93 to 3.72] | -3.85 [-6.25 to -1.44]
Statistical Analysis 1: Comparison: Placebo (Non-diabetic Obesity) vs PF-06882961 200 mg BID (Non-diabetic Obesity); Test type: Superiority; p = 0.0826, Mixed Models Analysis — 1-Sided; MMRM; Mean Difference (Final Values) = -3.74, 90% CI 2-sided [-8.23 to 0.75] — Test = PF-06882961 Reference = Placebo

ADVERSE EVENTS:
Time Frame: Baseline through follow-up (Day 112-119).
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Placebo (T2DM) | Placebo (Non-diabetic Obesity) | PF-06882961 80 mg BID Low, Slow (T2DM) | PF-06882961 80 mg BID High, Slow (T2DM) | PF-06882961 120 mg BID Low, Fast (T2DM) | PF-06882961 120 mg BID High, Fast (T2DM) | PF-06882961 200 mg BID (T2DM) | PF-06882961 200 mg BID (Non-diabetic Obesity)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6 | 0/20 | 0/22 | 0/22 | 0/22 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/20 | 0/22 | 0/22 | 0/22 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 8/16 | 4/6 | 11/20 | 13/22 | 14/22 | 14/22 | 14/21 | 18/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (T2DM) (N=16) | Placebo (Non-diabetic Obesity) (N=6) | PF-06882961 80 mg BID Low, Slow (T2DM) (N=20) | PF-06882961 80 mg BID High, Slow (T2DM) (N=22) | PF-06882961 120 mg BID Low, Fast (T2DM) (N=22) | PF-06882961 120 mg BID High, Fast (T2DM) (N=22) | PF-06882961 200 mg BID (T2DM) (N=21) | PF-06882961 200 mg BID (Non-diabetic Obesity) (N=22)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Pinguecula (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 2 | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 5 | 5 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 5 | 1 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 4 | 5 | 6 | 8 | 10 | 13
Vomiting (Gastrointestinal disorders) | 2 | 0 | 5 | 4 | 6 | 9 | 6 | 10
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Pre-existing condition improved (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infected bite (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 4 | 1 | 4 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 0 | 3 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 1 | 2 | 2 | 0 | 4
Headache (Nervous system disorders) | 1 | 1 | 1 | 3 | 1 | 1 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT04617275/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT04617275/SAP_001.pdf